CLINICAL TRIAL: NCT00211094
Title: A Placebo-Controlled, Double-blind, Randomized, Parallel Study of the Efficacy and Safety of Dapoxetine HCl in the Treatment of Rapid Ejaculation
Brief Title: A Study of the Effectiveness and Safety of Dapoxetine in the Treatment of Men With Premature Ejaculation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006091
Record Dates: First submitted 2005-09-15; First posted 2005-09-21 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: Ejaculation
Keywords: dapoxetine; premature ejaculation; ejaculation; sexual dysfunction; orgasmic disorder; sexual intercourse
MeSH Terms: conditions — Premature Ejaculation; Sexual Dysfunction, Physiological; Sexual Dysfunctions, Psychological; Coitus | interventions — dapoxetine

INTERVENTIONS:
Drug: Dapoxetine

SUMMARY:
The primary purpose of the study is to demonstrate that dapoxetine can prolong intravaginal ejaculatory latency time (IELT) compared with placebo in men with premature ejaculation (PE).

DETAILED DESCRIPTION:
One form of male sexual dysfunction is premature ejaculation (PE), which is also referred to as rapid ejaculation (RE). The study consists of 2 phases: pre-randomization phase (a screening visit and a 2-week baseline period); 12-week double-blind treatment phase during which patients will receive one of 2 doses of dapoxetine or placebo for use on an "as-needed" basis. The total duration of the study is approximately 14 weeks. Assessments of effectiveness include the average intravaginal ejaculatory latency time (as measured by stopwatch) during sexual intercourse, during the treatment period; control over ejaculation, participant and partner satisfaction with sexual intercourse, participant overall impression of change and severity of symptoms, based on questions asked at monthly intervals through the treatment phase. Safety assessments include the incidence, severity, and type of adverse events during the study, ECGs, as well as laboratory tests. At the end of the baseline period, patients from selected study centers will undergo blood sampling and ECG monitoring before and after the first dose of study medication. The study hypothesis is that treatment for 12 weeks with dapoxetine prolongs intravaginal ejaculatory latency time, compared with placebo, in men with PE. Oral tablets of dapoxetine (30 milligrams [mg] or 60mg) or placebo taken as needed during 12 weeks of treatment. No more than 1 dose within a 24-hour period.

ELIGIBILITY:
Inclusion Criteria:

* Patient is in a stable, monogamous sexual relationship with the same woman for at least 6 months and plans to maintain this relationship for the duration of the study
* history of premature ejaculation in the 6 months before study initiation not due to distress, interpersonal difficulty or medication withdrawal
* history of intravaginal ejaculatory latency time (IELT) of < = 2 minutes in at least 3 out of 4 events
* blood pressure < = 180/100 mmHg at screening and end of baseline
* patient and partner must agree to attempt sexual intercourse at minimum intervals specified in the protocol
* patient's partner must have a negative urine pregnancy test at time of screening

Exclusion Criteria:

* Not taken dapoxetine in a previous investigational drug study
* not using other forms of therapy for treatment of PE (behavioral therapy or medications applied to the skin)
* no history of any medical events that are associated with the development of PE
* not taken another investigational drug within 1 month
* no history of seizures or major psychiatric disorder such as depression or schizophrenia
* no alcohol abuse and dependence
* no known allergy or hypersensitivity to dapoxetine or other selective serotonin reuptake inhibitors (SSRIs)
* no partners with decreased interest in or painful intercourse or other forms of sexual dysfunction

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1320 (Actual)
Dates: Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Average intravaginal ejaculatory latency time (IELT), as measured by stopwatch, during sexual intercourse at the end of the treatment period (Week 12) for both doses of dapoxetine

SECONDARY OUTCOMES:
Control over ejaculation, satisfaction with sexual intercourse, and severity of symptom impressions, based on questions asked at monthly intervals through Week 12; incidence, severity, and type of adverse events throughout study; medication helpfulness

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA

REFERENCES:
- [Result] Pryor JL, Althof SE, Steidle C, Rosen RC, Hellstrom WJ, Shabsigh R, Miloslavsky M, Kell S; Dapoxetine Study Group. Efficacy and tolerability of dapoxetine in treatment of premature ejaculation: an integrated analysis of two double-blind, randomised controlled trials. Lancet. 2006 Sep 9;368(9539):929-37. doi: 10.1016/S0140-6736(06)69373-2. PMID 16962882
- [Derived] McMahon CG, Althof SE, Kaufman JM, Buvat J, Levine SB, Aquilina JW, Tesfaye F, Rothman M, Rivas DA, Porst H. Efficacy and safety of dapoxetine for the treatment of premature ejaculation: integrated analysis of results from five phase 3 trials. J Sex Med. 2011 Feb;8(2):524-39. doi: 10.1111/j.1743-6109.2010.02097.x. Epub 2010 Nov 8. PMID 21059176